CLINICAL TRIAL: NCT05225701
Title: Acceptability, Efficacy and Moderators of Clinical Change of a Transdiagnostic Guided Internet-Delivered Intervention for Emotional, Trauma and Stress-Related Disorders in the Mexican Population: Randomized Controlled Trial
Brief Title: Efficacy of a Transdiagnostic Guided Internet-Delivered Intervention for Emotional, Trauma and Stress-Related Disorders.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Anabel De La Rosa Gomez, Principal Investigator, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNAM_FESI_CONACYT_1401
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Emotional Disorder; Trauma and Stressor Related Disorders; Anxiety Disorders; Depression
Keywords: Transdiagnostic intervention; Guided Internet-Delivered intervention; Mexican population; Adults; Telepsychology; Internet-based treatment
MeSH Terms: conditions — Trauma and Stressor Related Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: A randomized controlled study will be carried out, in accordance with the guidelines set out in the consort (http://www.consort-statement.org) and CONSORT E-Health (https://www.jmir.org/2011/4/e126/). An experimental design will be used between subjects with three independent groups, with intrasubject measurements in four evaluation moments: pretest, posttest, follow-up at 3, 6 and 12 months (Solomon et al. ,2009). Participants will be randomly assigned to one of three conditions: a) Transdiagnostic guided internet-delivered intervention with synchronous assistance; b) Transdiagnostic self-guided internet-delivered intervention; c) waiting list.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded: The initial interview by the evaluator will be recorded and the video/audio will be shared with an independent evaluator who does not know the case for evaluation. Once the evaluation is completed, users will be randomly assigned to one of the study conditions. The randomization will be carried out by an independent researcher through the random.stg software in a 1: 1: 1 ratio by saturation of blocks of 12 per condition. The coordinator will inform the participant if he / she will participate in the study and, depending on the characteristics of the study design condition, he / she will be assigned to the self-guided/ guided intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transdiagnostic guided internet-delivered intervention with synchronous assistance (Experimental): Self-applied treatment web system based on transdiagnostic approach for emotional and stress and trauma-derived disorders. The system will contain seven modules. The duration of the intervention program may vary between users; however, the participant will have access permits for a maximum period of 12 weeks. In order to monitor the participant's progress, each user will be assigned an advisor who will be health personnel (psychologists, social workers, and gerontologists) to get an a weekly personalized synchronous assistance and psychological counseling.
  Interventions: Behavioral: Transdiagnostic guided internet-delivered intervention with synchronous assistance
- Transdiagnostic self-guided internet-delivered intervention (Active Comparator): Self-applied treatment web system based on transdiagnostic approach for emotional and stress and trauma-derived disorders. The system will contain seven modules. The duration of the intervention program may vary between users; however, the participant will have access permits for a maximum period of 12 weeks. All modules are sequential, allowing the user to go step by step. This arm does not have personalized online assistance.
  Interventions: Behavioral: Transdiagnostic self-guided internet-delivered intervention
- waiting list (No Intervention): Participants on the waiting list will be assigned to the intervention after 2 months after randomization and will join the Transdiagnostic guided internet-delivered intervention with synchronous assistance.

INTERVENTIONS:
Behavioral: Transdiagnostic guided internet-delivered intervention with synchronous assistance — Self-applied treatment web system based on transdiagnostic approach for emotional and stress and trauma-derived disorders. The system will contain seven modules: Module 0. Pre-evaluation; Module 1. Psychoeducation and motivation for change; Module 2. Emotional Coping Skills; Module 3. Acceptance and awareness-raising skills focused on the present moment; Module 4. Cognitive coping skills; Module 5. Behavioral coping skills; Module 6. Achievements, maintenance and prevention of relapses; Module 7. Post-evaluation. Each user will be assigned an advisor who will be health personnel (psychologists, social workers, and gerontologists). The function of the psychological advisor is to motivate, guide and listen to the doubts and comments of each participant by providing a weekly session of one hour in individual online format, in addition to the review of the module in platform in self-suggestive format.
  Arms: Transdiagnostic guided internet-delivered intervention with synchronous assistance
Behavioral: Transdiagnostic self-guided internet-delivered intervention — Self-applied treatment web system based on transdiagnostic approach for emotional and stress and trauma-derived disorders. The system will contain seven modules: Module 0. Pre-evaluation; Module 1. Psychoeducation and motivation for change; Module 2. Emotional Coping Skills; Module 3. Acceptance and awareness-raising skills focused on the present moment; Module 4. Cognitive coping skills; Module 5. Behavioral coping skills; Module 6. Achievements, maintenance and prevention of relapses; Module 7. Post-evaluation. Each module will include exercises and tasks for the practice of each technique. Automatic emails with notifications will be sent to access the program when participants have not entered in the last 15 days.
  Arms: Transdiagnostic self-guided internet-delivered intervention

SUMMARY:
Emotional, trauma and stress-related disorders show high incidence, prevalence, morbidity, and comorbidity rates in Mexico. In recent decades, research findings indicate that cognitive behavioral interventions, from a disorder-specific perspective, are the effective front-line treatment for anxiety and depression care. However, these treatments are not often used. The reasons for this are: limited access and low availability to effective interventions; a minority of people actively seek psychological care because of their own distress condition, fearing social stigma, because of geographical reasons that separate them from health centers, because of time, preference for other treatment or self-help, for the high cost of treatment, which makes it inaccessible and unaffordable to both, the user, and the public health system. It has also been stated that the comorbidity between mental disorders, as well as the gap between research findings and clinical practice could influence the poor dissemination of effective treatments, resulting in a lack of up-to-date professionals providing relevant interventions. This has motivated the practice of some studies aimed at knowing the moderating, mediating variables and psychological mechanisms that improve the process of clinical change. Emotional deregulation of negative affection has been found to be a moderating factor and/or mediation in addressing emotional disorders from a transdiagnostic perspective, aimed at two or more specific disorders. In this way, transdiagnostic treatments could help overcome the drawbacks related to comorbidity between disorders. However, technological advancement has created alternatives for psychological assistance, highlighting the possibilities offered by technologies since Internet-supported interventions have been empirically tested for effectiveness, efficiency and this efficiency can be key to ensuring access to those who are inaccessible. Thus, the study aims to identify the indicators of efficacy, acceptability, and moderation of clinical change of a transdiagnostic intervention through a telepsychology platform for the treatment of emotional disorders and derived from stress and trauma.

DETAILED DESCRIPTION:
Individuals suffering from depression are more likely to develop comorbidity with other mental disorders, an estimated 53% have concurrent symptomatology with some anxiety disorder (Weisel et al., 2018). Stress and traumatic events are among the most relevant causes, between 60% and 80%, contributing to the etiology of emotional disorders. Depression and anxiety have also been deemed to create a condition of greater disability by increasing the severity and chronicity rate of psychological discomfort and is associated with increased mortality in medical conditions such as heart disease, chronic-degenerative or psychiatric conditions (Berenzon et al., 2013). In Mexico, one in four people between the age of 18 and 65 has suffered an emotional disorder at some point in their lives, but only one in five of those with it receive treatment and the time to receive care in a health center ranges from 4 to 20 years depending on the reason for consultation (Berenzon et al., 2013).

In recent decades, cognitive behavioral interventions, from a disorder-specific perspective, constitute an effective and first-line treatment for anxiety and depression care (Cuijpers et al. 2014; Kazdin, 2016); They highlight: a) exposure therapy; b) anxiety management techniques; and c) cognitive therapy, however, however they are not often used (Mohr et al., 2010). In this regard, a number of reasons have been noted explaining limited access and low availability to effective interventions. A minority of people actively seek psychological care because of their own condition of emotional discomfort, fearing social stigma, because of geographical reasons that separate them from health centers, because of reasons of time, preference for other treatment or self-help, because of the high cost of psychological support, which makes it inaccessible and unaffordable to both, the user and the public health system (Berenzon et al., 2013). It has also been argued that the comorbidity between mental disorders, as well as the gap between research findings and clinical practice could influence the poor dissemination of effective treatments; resulting in a lack of up-to-date professionals providing relevant interventions (Holmes, Craske & Graybiel, 2014). In the same line, Kazdin and Blase (2011) mention that, despite advances in research, mental health professionals have been unsuccessful in reducing the incidence and prevalence of emotional disorders. This has motivated studies aimed at knowing the moderating, mediating variables and psychological mechanisms that improve the process of clinical change (Ebert et al., 2018). In addition, the need has been raised to implement innovative solutions that contribute to the dissemination of effective treatments for the care of emotional disorders( Kazdín & Rabbitt, 2016).

Faced with this problem, psychological rehabilitation of people diagnosed with depression and anxiety has been found to be mediated by the primary assessment of the event that can be perceived as threat, challenge, or benefit; estimation of control over adverse or stressful stimulus and the resources available to deal with the situation (Folkman & Moskowitz, 2007). In particular, emotional deregulation of negative affection is a study factor that is providing relevant data for better understanding and approaching emotional disorders from a transdiagnostic perspective, a term coined from a dimensional conception to designate effective treatments targeting two or more specific disorders (Hernández et al., 2011).

This has crucial implications for the possible diagnosis of emotional disorders, since, from a dimensional perspective, consideration of the causes and coping resources that the person has and not only the count of prescribed grouped symptoms takes on relevance. The degree of intensity and effects on the day-to-day functioning of the person are also taken into account. For treatment purposes, it addresses common or shared risk factors between disorders (e.g. emotional disorders), including underlying mechanisms, psychological (cognitive, behavioral and physiological) processes linked to explanatory variables and maintenance of overlapping symptoms (attentional biases, negative thinking, avoidance, etc.), appealing to a convergent and integrative scientific approach (Sandin, 2014). Thus, transdiagnostic treatments could help overcome the disadvantages related to comorbidity between disorders and thus make way for a new generation of emotion-focused treatments (Hernández et al., 2011). In this regard, Barlow, Allen and Choate (2004) return to the tripartite theory of emotion (Clark & Watson, 1991) and propose a unified cognitive-behavioral transdiagnosis protocol for the treatment of emotional disorders with an emphasis on emotional regulation.

On the one hand, there is evidence of effective transdiagnostic interventions for the treatment of emotional disorders that help overcome the disadvantages related to comorbidity between disorders; and on the other hand, the benefits shown by interventions provided over the Internet and mobile applications by allowing: (1) accessibility: easy access anytime and from anywhere over the Internet, (2) flexibility: the intervention adapts to the participant's pace and the consultation of resources and materials can be asynchronous, (3) customization: the intervention can be adapted to the specific needs of the user, (4) availability of treatment: it allows to bring psychological care to people who need it regardless of distance, which is an alternative when it is not possible to access face-to-face mental health services. In addition, (5) scalability, as it can increase coverage and improve care as technology advances (Díaz-García, 2017; Weisel et al., 2018). Therefore, transdiagnostic interventions focused on the emotion provided online involve enhancing the scope and impact of psychological treatment programs for anxiety and depression (Titov et al., 2013).

While there is evidence of effectiveness, aimed at knowing the impact of the outcome of treatment, other relevant aspects that has not been sufficiently explored are the risk and/or protection factors that cause moderation and mediation effects with respect to the results obtained in treatments (Graaf et al., 2002) for example, to know the profiles that benefit most from interventions (Brookes et al., 2004; Kessler et al., 2017). Identifying variables that moderate or mediate the impact of treatment is important because it could support understanding the heterogeneity of the results. Evidence of the effectiveness of preventive and/or remedial interventions over the Internet in the context of public health for the reduction of the incidence of depressive and anxious symptomatology is still low; the latest systematic review identified seven uncontrolled clinical studies that evaluated the effect of internet-mediated interventions with positive results (Ebert et al., 2017). However, only one clinical study aimed at preventing general anxiety was found that did not produce significant results (Christensen et al., 2014). While three studies managed to reduce the incidence of depression (Buntrock et al., 2016; Dear et al., 2016). In the study conducted by Dear et al. (2016) reported that self-applied internet-guided intervention decreased depressive symptomatology in a group of adults and managed to reduce the risk of chronic depression by 39% per follow-up year. Recent research on the effectiveness of self-applied interventions via the Internet with and without the support of a trained psychologist has indicated that fully self-applied technology-mediated treatments show fewer rates of improvement compared to those who did have synchronous support with a therapist (Richards & Richardson, 2012). Other studies that have researched the influence of support or guidance during self-applied internet-based interventions have reported that participants who received weekly support significantly improved in reducing depression compared to a waiting list group, while participants who did not receive support did not show significant improvement (Kleiboer et al., 2015). However, some authors propose that the differences in results obtained between guided and non-guided interventions are small or non-existent (Mira et al., 2017). This aspect is relevant for assessing the efficiency of interventions provided with technology, as they could benefit more people who need it with effective results. In general, the research findings mentioned are promising; however, it is also important to note that most studies have been conducted in developed contries, so it is necessary to know the results in controlled studies in the Mexican context and culture and with larger samples to reach stronger conclusions regarding the effectiveness, efficacy and efficiency of transdiagnostic interventions via the Internet for the care of emotional disorders. In addition, it is necessary to investigate what are the suitable applications of the technology, whether or not there is a significant benefit using this technology compared to other strategies that are currently available, and what factors can contribute to these effects (Quero et al., 2012).

In Mexico, research in this area is incipient, emphasizing the need to go beyond traditional face-to-face interventions and to design new intervention strategies. In this regard, the possibilities offered by technologies are highlighted since Internet-supported interventions have been empirically tested to achieve effectiveness and efficiency/cost-benefit and can be key to ensuring access to those who are inaccessible. Thus, in consistency with the National Health Plan, this study aims to respond to this national problem through the evaluation of the effectiveness and moderators of a transdiagnostic intervention for emotional disorders through a telepsychology system.

ELIGIBILITY:
Inclusion Criteria:

a) be of legal age; b) voluntarily participate in the study; c) meet diagnostic criteria for emotional disorders (anxiety or depression) in accordance with the International Neuropsychiatric Interview- Mini, version 5.0 (Sheehan et al., 2006), and show a score ≤ 25 in Beck's Anxiety Depression Inventory (Beck & Steer,1990) and/or ≤ 30 in the Beck-BDI-II Depression Inventory (Beck, Steer & Brown, 1996); d) have access to computer equipment with an Internet connection; e) have a valid email address; f) have basic digital skills in the use of an operating system and internet browsing.

Exclusion Criteria:

a) psychotic disorder; b) alcohol and drug abuse; c) have active suicidal ideation; d) medical condition whose severity or characteristics prevent the intervention; e) be receiving psychological and/or pharmacological treatment during the study.

Elimination criteria :

a) not accepting the conditions of informed consent and b) absence on web or mobile platform for more than 15 days or having missed two consecutive sessions of synchronous treatment sessions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in the score of Beck Anxiety Inventory | 9 weeks
  Beck Anxiety Inventory (BAI , Beck & Steer, 1990). The BAI is a 21-item self-report measure of the severity of common affective, cognitive, and somatic symptoms of anxiety. Items have four response options ranging from 0 "not at all" to 3 "severely". The cut-off points are: 0-5 minimal anxiety, 6-15 mild anxiety, 16-30 moderate anxiety and 31-63 severe anxiety. High internal consistency and adequate construct validity, divergent and convergent for the Mexican version has been documented (Cronbach's alpha = .83) (Robles et al., 2001).
Decrease in the score of Beck Depression Inventory | 9 weeks
  Beck Depression Inventory (BDI-II; Beck, Steer & Brown, 1996). It consists of 21 items that fundamentally evaluate the clinical symptoms of melancholy and the intrusive thoughts present in depression. Cronbach's alpha for version II (= .87-.92). Each statement has four response options that reflect increasing symptom frequency or severity. Total scores can range from 0-63 with the following cut-offs points: 0-13 minimally depressed, 14-19 mildly depressed, 20-28 moderately depressed, and 29-63 severely depressed.
Decrease in the score of Post-Traumatic Stress Disorder Checklist | 9 weeks
  This instrument describes the symptoms of post-traumatic stress taking into consideration the diagnostic criteria of activation, alterations, avoidance and reexperimentation. It has 20 items that are scored on a Likert-type scale that goes from 0 (not at all) to 4 (totally). In its adaptation to the Mexican population, the psychometric properties of the scale show adequate internal consistency with an alpha of .97, as well as an appropriate convergent validity (rs = .58 to .88; Durón-Figueroa et al., 2019). Items are scored on a Likert scale ranging from 0 to 4, where higher scores indicate more pronounced PTSD symptoms. A cut-off score of 33 was suggested to have a partial diagnosis of PTSD.
Decrease in the score of Scale of Difficulties in Emotional Regulation | 9 weeks
  Scale of Difficulties in Emotional Regulation (DERS; Gratz & Roemer, 2004). It is a self-applied instrument that measures two dimensions through 15 items, emotional regulation strategies and awareness of emotions. The version validated in Mexican population by De la Rosa et al. (2021), presents a Cronbach's Alpha valued between .84 - .74.
Decrease frequency, severity and avoidance of anxiety | 9 weeks
  General Anxiety and the Impairment Severity Scale (OASIS) (Norman et al., 2011). It consists of 5 questions with a scale of 0 to 4, which measures frequency, severity and avoidance of anxiety in different fields: work / academic interference / family, and deterioration of social and daily life. It has good internal consistency (α = 0.80) and test-retest reliability (k = 0.82). The Spanish version confirmed the factorial structure, reliability and validity data obtained by the original authors: internal consistency in both populations, in general and clinical (α = 0.86) and test-fail reliability (k = 0.84) (Mira et al., 2015).
Decrease frequency and severity of depression | 9 weeks
  General Depression and the Impairment Gravity Scale (ODSIS)(Bentley et al., 2014). This scale evaluates experiences related to depression. It consists of five items with different answer options ranging from 0 to 4 for each item. It measures the frequency and severity of depression, as well as the level of avoidance to work/academic/home interference, and social life. In the Spanish version, the internal consistency has proven to be excellent, with a Cronbach alpha between 0.91 and 0.94 and a good convergent and discriminatory validity (González-Robles et al., 2015).

SECONDARY OUTCOMES:
Increase the level of acceptance and satisfaction of psychological treatment | 9 weeks
  Questionnaire with four questions that report the level of satisfaction with the treatment, if you would recommend the treatment to a friend or relative, is the treatment considered useful for your case and if you think that the treatment was difficult to handle or aversive.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel García Flores, PhD, Study Chair — Technological Institute of Sonora, Department of Psychology; Enrique Berra Ruiz, PhD, Study Chair — Autonomous University of Baja California, Faculty of Health Sciences / Psychology; Esteban E Esquivel Santoveña, PhD, Study Chair — Department of Social Sciences, Autonomous University of Ciudad Juárez (UACJ); Paulina Arenas Landgrave, PhD, Study Chair — Faculty of Psychology, National Autonomous University of Mexico; Rocío Silvestre Ramírez, MD, Study Chair — Comprehensive Center for Mental Health Tzompantepec, Secretary of Health Tlaxcala; Rosa O Castellanos Vargas, MA, Study Chair — Health Sciences, Autonomous University of Ciudad Juárez (UACJ); Alicia I Flores Elvira, MA, Study Chair — Faculty of Higher Studies Iztacala, National Autonomous University of Mexico; Alejandro Domínguez-Rodríguez, PhD, Study Chair — International University of Valencia; Carolina Santillán Torrres Torija, PhD, Study Chair — Faculty of Higher Studies Iztacala, National Autonomous University of Mexico
Locations (6):
- Mexico (6):
  - Autonomous University of Ciudad Juarez, Ciudad Juárez, Chihuahua
  - Autonomous University of Baja California, Tijuana, Estado de Baja California
  - Instituto Tecnológico de Sonora, Ciudad Obregón, Sonora
  - Faculty of Higher Studies Iztacala, National Autonomous University of Mexico, Tlalnepantla, State of Mexico, Mexico
  - Comprehensive Mental Health Center, Ministry of Health of Tlaxcala, Santa Ana Chiautempan, Tlaxcala
  - Faculty of Psychology, National Autonomous University of Mexico, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a open server of the journal(s) that we will publish the articles that will be the result of this study. The informed consent is already shared in the register of clinical trials.
Supporting Information: Study Protocol, ICF
Time Frame: This data will be available in december 2023 and it will be available for 5 years. It will be shared in the databases of the journal where the article(s) will be published.
Access Criteria: Open access saving personal and sensitive data of the participants.

REFERENCES:
- [Background] Andersson G. Internet-Delivered Psychological Treatments. Annu Rev Clin Psychol. 2016;12:157-79. doi: 10.1146/annurev-clinpsy-021815-093006. Epub 2015 Dec 11. PMID 26652054
- [Background] Barlow DH, Allen LB, Choate ML. Toward a Unified Treatment for Emotional Disorders - Republished Article. Behav Ther. 2016 Nov;47(6):838-853. doi: 10.1016/j.beth.2016.11.005. Epub 2016 Nov 10. PMID 27993336
- [Background] Health Quality Ontario. Internet-Delivered Cognitive Behavioural Therapy for Major Depression and Anxiety Disorders: A Health Technology Assessment. Ont Health Technol Assess Ser. 2019 Feb 19;19(6):1-199. eCollection 2019. PMID 30873251
- [Background] Dominguez-Rodriguez A, De La Rosa-Gomez A, Hernandez Jimenez MJ, Arenas-Landgrave P, Martinez-Luna SC, Alvarez Silva J, Garcia Hernandez JE, Arzola-Sanchez C, Acosta Guzman V. A Self-Administered Multicomponent Web-Based Mental Health Intervention for the Mexican Population During the COVID-19 Pandemic: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Nov 16;9(11):e23117. doi: 10.2196/23117. PMID 33196449
- [Background] Dominguez-Rodriguez A, Martinez-Luna SC, Hernandez Jimenez MJ, De La Rosa-Gomez A, Arenas-Landgrave P, Esquivel Santovena EE, Arzola-Sanchez C, Alvarez Silva J, Solis Nicolas AM, Colmenero Guadian AM, Ramirez-Martinez FR, Vargas ROC. A Self-Applied Multi-Component Psychological Online Intervention Based on UX, for the Prevention of Complicated Grief Disorder in the Mexican Population During the COVID-19 Outbreak: Protocol of a Randomized Clinical Trial. Front Psychol. 2021 Mar 29;12:644782. doi: 10.3389/fpsyg.2021.644782. eCollection 2021. PMID 33854466
- [Background] Ontario Health (Quality). Internet-Delivered Cognitive Behavioural Therapy for Post-traumatic Stress Disorder or Acute Stress Disorder: A Health Technology Assessment. Ont Health Technol Assess Ser. 2021 Jun 1;21(9):1-120. eCollection 2021. PMID 34527087
- [Derived] de la Rosa-Gomez A, Flores-Plata LA, Esquivel-Santovena EE, Santillan Torres Torija C, Garcia-Flores R, Dominguez-Rodriguez A, Arenas-Landgrave P, Castellanos-Vargas RO, Berra-Ruiz E, Silvestre-Ramirez R, Miranda-Diaz GA, Diaz-Sosa DM, Hernandez-Posadas A, Flores-Elvira AI, Valencia PD, Vazquez-Sanchez MF. Efficacy of a transdiagnostic guided internet-delivered intervention for emotional, trauma and stress-related disorders in Mexican population: study protocol for a randomized controlled trial. BMC Psychiatry. 2022 Aug 9;22(1):537. doi: 10.1186/s12888-022-04132-6. PMID 35941557

DOCUMENTS (1):
  • Informed Consent Form (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05225701/ICF_000.pdf